CLINICAL TRIAL: NCT01265186
Title: Evaluation of Sedation in Newborns - a Prospective, Controlled, Observer Blinded Clinical Trial in 67 Patients
Brief Title: Evaluation of Sedation in Newborns
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Philipp Deindl, Medical University of Vienna
Other Study IDs: 704/2010
Record Dates: First submitted 2010-12-22; First posted 2010-12-23 (Estimated); Last update posted 2010-12-23 (Estimated); Status verified 2010-12

CONDITIONS: Sedation
Keywords: Sedation; BIS; aEEG; Neonatal Pain and Sedation Scale; neonate; newborn
MeSH Terms: interventions — Consciousness Monitors

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Ventilated term newborns: Ventilated newborns with a corrected gestational age ≧ 37 weeks of gestation until the 28th day of life respectively ≦ 44 weeks of gestation
  Interventions: Device: Bispectral Index; Device: Amplitude-integrated EEG
- Control group: healthy term newborns: Control group: healthy newborns with a corrected gestational age ≧ 37 weeks of gestation until the 28th day of life respectively ≦ 44 weeks of gestation
  Interventions: Device: Bispectral Index; Device: Amplitude-integrated EEG

INTERVENTIONS:
Device: Bispectral Index — The Bispectral-Index is continuously recorded for up to 72 hours in the group of ventilated newborns. Every 15 minutes, a value that was generated by averaging the BIS values of the last 15 minutes will be recorded (automatically calculated by the software of the readout device). The Bispectral-Index is continuously recorded for a minimum of 4 hours in the controls.
  Other Names: BIS VISTA™ Monitoring System, Covidien
Device: Amplitude-integrated EEG — A aEEG is recorded once daily for a minimum of four hours in the group of ventilated newborns. In Controls an aEEG is recorded once for a minimum of four hours.
  Other Names: The Olympic CFM 6000

SUMMARY:
Neonates treated on Neonatal Intensive Care Units are often critically ill, subject to numerous painful procedures and often dependent on mechanical ventilation. Mechanical ventilation as well as painful conditions require a sufficient analgesia and or an accurately regulated sedation. Newborns incapable of self-report are therefore dependent on the assessment of the infants level of pain and sedation by the treating team.

The aim of this prospective, controlled, observer-blinded clinical trial is to compare the performance of two EEG based methods and a clinical sedation scale to measure the level of sedation in neonates. The Bispectral-Index (BIS) and the amplitude-integrated EEG (aEEG) are compared with the Neonatal Pain and Sedation Scale (N-PASS). We hypothesize a correlation between the clinical sedation score (N-PASS), the bispectral index (BIS) and the amplitude-integrated EEG (aEEG). Fifty-two mechanically ventilated term neonates and fifteen control patients are enrolled and observed for up to 72h.

ELIGIBILITY:
Inclusion Criteria:

* newborns with a corrected gestational age ≧ 37 and ≦ 44 weeks of gestation

Exclusion Criteria:

* congenital malformations
* chromosomal aberrations
* brain abnormalities
* severe cerebral hemorrhage (grade III-IV)
* cystic periventricular leukomalacia
* infections of the central nervous system

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Ventilated term newborns with or without pharmacological sedation/analgesia
Sampling Method: Probability Sample
Enrollment: 67 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Correlation between clinical sedation score (N-PASS) and the bispectral index (BIS) and the amplitude-integrated EEG (aEEG) | 72 hours
  The BIS-Monitoring is continuously recorded for up to 72 hours.A aEEG is recorded once daily for a minimum of four hours. aEEG and BIS are derived continuously for two head electrodes. Every 3-4 hours the N-PASS is evaluated by a nurse and recorded in the patient documentation system.

SECONDARY OUTCOMES:
Differences of the values of the BIS, the aEEG and the sedation scores in the group of mechanically ventilated / sedated newborns and the group of non-ventilated /non-sedated neonates | 72 hours
  Comparison of sedation levels between the two groups
Relationship between daily doses of sedatives / analgesics and sedation levels | 72 hours
  Relationship between daily doses of sedatives / analgesics and sedation levels

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatrics and Adolescent Medicine, Division of Neonatology, Medical University of Vienna, Vienna, Austria